CLINICAL TRIAL: NCT03081585
Title: Integration of Homeostatic Signaling and Food Reward Processing in the Human Brain
Brief Title: Food Reward Processing in the Human Brain
Status: Completed | Type: Observational
Sponsor: University of Heidelberg Medical Center (Other)
Responsible Party: Principal Investigator, Joe Simon, Principal Investigator, University of Heidelberg Medical Center
Other Study IDs: NSM
Record Dates: First submitted 2017-03-10; First posted 2017-03-16 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Healthy
Keywords: fmri; neuronal reward processing; hormonal satiety signalling; fasting
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Controls: Normal weight, healthy female participants
  Interventions: Behavioral: Satiety State

INTERVENTIONS:
Behavioral: Satiety State — Participants were scanned twice: once after a meal and once after fasting for 24 hours

SUMMARY:
The aim of this study is to investigate the influence of different metabolic states and hormonal satiety signalling on responses in neural reward networks.

DETAILED DESCRIPTION:
Given the rapid development of obesity world-wide, a better understanding of the interaction between the encoding of food reward in mesocorticolimbic reward pathways and homeostatic energy regulation is of paramount importance for the development of new treatment strategies. Healthy participants will undergo functional magnetic resonance imaging while performing a task distinguishing between the anticipation and the receipt of either food or monetary reward. Every participant will be scanned twice in a counterbalanced fashion, both during a state of hunger (after 24-hours fasting) and satiety. Blood samples will be collected to assess hormonal satiety signalling. We hope to provide new insights into the neurobiological underpinnings of motivational processing and hedonic evaluation of food reward.

ELIGIBILITY:
Inclusion Criteria:

* BMI <25 kg/m² and >18.5 kg/m²
* no lifetime or current medical illness that could potentially affect appetite or body weight
* right-handedness
* normal or corrected-to-normal vision

Exclusion Criteria:

* history of head injury or surgery
* history of neurological disorder
* severe psychiatric disorder (psychosis, bipolar disorder, substance abuse)
* smoking
* borderline personality disorder
* current psychotropic medication
* inability to undergo fMRI scanning (e.g. metallic implants, claustrophobia, Pacemakers)
* pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy normal weight female participants
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2015-06-09 (Actual); Primary Completion 2016-06-10 (Actual); Study Completion 2016-06-10 (Actual)

PRIMARY OUTCOMES:
Experimental fMRI task (incentive delay task) | 22 min.
  Participants were expecting food and monetary related reward, after a correct response to a simple task they received either food or monetary related reward.
Resting state brain activity using functional magnetic resonance imaging | 5 min.
  Functional brain imaging will be employed to assess functional connectivity in reward related brain networks.

SECONDARY OUTCOMES:
Analysis of hormonal satiety signaling | 30 min. before scanning
  Blood is collected for the measurement of peripheral ghrelin. One blood sample at the start of the experiment will be collected.
Self-report questionnaire regarding eating behavior (Dutch Eating Behavior Questionnaire) | 30 min.
  Psychometric tests will be employed to assess eating behavior and eating disorder psychopathology (using the Dutch Eating Behavior Questionnaire).

CONTACTS AND LOCATIONS:
Overall Officials: Joe Simon, Dr. Dipl. Psych., Principal Investigator — University Hospital Heidelberg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Simon JJ, Wetzel A, Sinno MH, Skunde M, Bendszus M, Preissl H, Enck P, Herzog W, Friederich HC. Integration of homeostatic signaling and food reward processing in the human brain. JCI Insight. 2017 Aug 3;2(15):e92970. doi: 10.1172/jci.insight.92970. eCollection 2017 Aug 3. PMID 28768906